CLINICAL TRIAL: NCT00570713
Title: A Phase 2 Randomized, Placebo-controlled, Double-blind Study of the Efficacy of MORAb-009 in Combination With Gemcitabine in Patients With Advanced Pancreatic Cancer.
Brief Title: An Efficacy Study of MORAb-009 in Subjects With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MORAb-009-002
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Results first posted 2012-03-27 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — amatuximab; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MORAb-009 (Experimental): MORAb-009 plus gemcitabine ('MORAb-009'): MORAb-009 was administered at 5 mg/kg on Day 1 of Weeks 1 through 7 during the first cycle and on Day 1 of Weeks 1 through 3 of subsequent cycles. Gemcitabine was administered by i.v. infusion at an initial dose of 1000 mg/m2 once weekly for up to 7 weeks (or until toxicity necessitated reducing or holding a dose), followed by a week of rest from treatment. Subsequent cycles consisted of infusions once weekly for 3 consecutive weeks, followed by a week of rest from treatment.
  Interventions: Drug: MORAb-009; Drug: Gemcitabine
- Placebo (Active Comparator): Placebo plus gemcitabine ('Placebo') Placebo was administered on Day 1 of Weeks 1 through 7 during the first cycle and on Day 1 of Weeks 1 through 3 of subsequent cycles. Gemcitabine was administered by i.v. infusion at an initial dose of 1000 mg/m2 once weekly for up to 7 weeks (or until toxicity necessitated reducing or holding a dose), followed by a week of rest from treatment. Subsequent cycles consisted of infusions once weekly for 3 consecutive weeks, followed by a week of rest from treatment.
  Interventions: Drug: Placebo; Drug: Gemcitabine

INTERVENTIONS:
Drug: MORAb-009 — Monoclonal antibody administered once weekly by intravenous injection.
  Arms: MORAb-009
Drug: Placebo — As per package insert.
  Arms: Placebo
Drug: Gemcitabine — Gemcitabine was administered by i.v. infusion at an initial dose of 1000 mg/m2 once weekly for up to 7 weeks (or until toxicity necessitated reducing or holding a dose), followed by a week of rest from treatment. Subsequent cycles consisted of infusions once weekly for 3 consecutive weeks, followed by a week of rest from treatment.

SUMMARY:
The purpose of this study is to investigate the activity of MORAb-009 when added to a standard regimen of gemcitabine in patients with previously untreated unresectable stage 3 or 4 pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects, ≥ 18 years of age, with cytologically or histologically confirmed diagnosis of pancreatic adenocarcinoma.
2. Must have measurable disease, as defined by RECIST or evaluable by clinical signs/symptoms (e.g. ascites, pleural effusion, or lesions of less than 2 cm) supported by biomarker, radiologic, or pathologic studies conducted within 4 weeks prior to study entry.
3. Must have unresectable disease and have received no prior chemotherapy or radiation therapy for their pancreatic cancer.
4. Karnofsky performance status of greater than or equal to 70 %.
5. Female subjects of childbearing potential and all male subjects must be surgically sterile or consent to use a medically acceptable method of contraception throughout the study period.
6. Other significant medical conditions must be well-controlled and stable in the opinion of the investigator for at least 30 days prior to Study Day 1.
7. Laboratory and clinical results within the 2 weeks prior to Study Day 1 as follows:

   Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L Hemoglobin ≥ 9 g/dL Serum bilirubin ≤ 2.0 mg/dL Aspartate transaminase (AST)* ≤ 5 x upper limit of normal (ULN) Alanine transaminase (ALT)* ≤ 5 x ULN Alkaline phosphatase* ≤ 5 x ULN Serum creatinine ≤ 2.0 mg/dL Stenting to reduce liver functions to qualifying levels is permitted.

   * Subjects with liver function abnormalities greater than the ULN are eligible only if in the opinion of the investigator they are due to disease obstruction of the bile ducts or metastatic disease.
8. Must be willing and able to provide written informed consent.

Exclusion Criteria:

1. Known central nervous system (CNS) tumor involvement.
2. Evidence of other active malignancy requiring treatment.
3. Clinically significant heart disease (e.g., congestive heart failure of New York Heart Association Class 3 or 4 angina not well controlled by medication, or myocardial infarction within 6 months).
4. Electrocardiogram (ECG) demonstrating clinically significant arrhythmias (Note: Subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia [SVT], are eligible).
5. Active serious systemic disease, including active bacterial or fungal infection.
6. Active viral hepatitis or symptomatic human immunodeficiency virus (HIV) infection.
7. Prior chemotherapy or radiation therapy for their pancreatic cancer.
8. Breast-feeding, pregnant, or likely to become pregnant during the study.
9. No other concurrent immunotherapy (e.g., immunosuppressants or chronic use of systemic corticosteroids with the exception that low-dose corticosteroids are allowed)
10. Known hypersensitivity to a monoclonal antibody or biologic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (26):
  - Moores UCSD Cancer Center, La Jolla, California
  - Southern California Permanente Medical Group, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente, Vallejo, California
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Connecticut Oncology & Hematology, Torrington, Connecticut
  - Palm Beach Institute of Hematology and Oncology, Boynton Beach, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Hematology Oncology Associates of the Palm Beaches, Lake Worth, Florida
  - Hematology-Oncology Associates of Illinois, LLC, Skokie, Illinois
  - Carle Clinic Assoc., Urbana, Illinois
  - University of Kansas Medical Center, Westwood, Kansas
  - Jayne Gurtler, MD, Laura Brinz, MD, & Angelo Russo, MD, Metairie, Louisiana
  - Providence Cancer Center, Oncology, Clinical Trials, Southfield, Michigan
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Arena Oncology Associates, P.C., Lake Success, New York
  - Hanover Medical Specialists, MD, Wilmington, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Arlington Cancer Center, Arlington, Texas
  - Baylor College of Medicine, Houston, Texas
  - South Texas Onocology Hemotology, PA, San Antonio, Texas
  - Providence Western Washington Oncology, Lacey, Washington
  - Medical College of Wisconsin Clinical Cancer Center, Milwaukee, Wisconsin
- Belgium (3):
  - Centre Hospitalier Jolimont-Lobbes, Haine-Saint-Paul, Hainaut
  - Services de gastro-entérologie et d'oncologie, CHC Saint-Joseph, Liège
  - AZ Sint Maarten - digestive oncology unit - campus, Mechelen
- Canada (4):
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - London Regional Cancer Program London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital - Montreal, Montreal, Quebec
- Germany (7):
  - Klinik fuer Tumorbiologie an der Albert-Ludwigs-Universität Freiburg, Freiburg im Breisgau, Baden Wurttemburg
  - Nationales Centrum für Tumorerkrankungen (NCT) Heidelberg, Universitätsklinikum Heidelberg, Heidelberg, Baden Wurttemburg
  - SLK-Kliniken Heilbronn GmbH, Medizinische Klinik III, Heilbronn, Baden Wurttemburg
  - Universitätsklinikum Ulm, Innere Medizin I, Ulm, Baden Wurttemburg
  - II. Medizinische Klinik des Klinikums rechts der Isar, München, Bavaria
  - Stadtische Kliniken Bielefeld-Mitte, Klinik fur Hamatologie und Onkologie, Bielefeld, North Rhine-Westphalia
  - Charité, Universitätsmedizin Berlin, Berlin
- Spain (5):
  - Hospital Madrid, Madrid, Madrid
  - Hospital Clinico Universitario San Carlos, Madrid, Madrid
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital 12 de Octubre, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a population of pancreatic cancer patients treated at investigational centers.
Groups:
- MORAb-009 Plus Gemcitabine ('MORAb-009'): MORAb-009 was administered at 5 mg/kg on Day 1 of Weeks 1 through 7 during the first cycle and on Day 1 of Weeks 1 through 3 of subsequent cycles. Gemcitabine was administered by i.v. infusion at an initial dose of 1000 mg/m2 once weekly for up to 7 weeks (or until toxicity necessitated reducing or holding a dose), followed by a week of rest from treatment. Subsequent cycles consisted of infusions once weekly for 3 consecutive weeks, followed by a week of rest from treatment.
- Placebo Plus Gemcitabine ('Placebo'): Placebo was administered on Day 1 of Weeks 1 through 7 during the first cycle and on Day 1 of Weeks 1 through 3 of subsequent cycles. Gemcitabine was administered by i.v. infusion at an initial dose of 1000 mg/m2 once weekly for up to 7 weeks (or until toxicity necessitated reducing or holding a dose), followed by a week of rest from treatment. Subsequent cycles consisted of infusions once weekly for 3 consecutive weeks, followed by a week of rest from treatment.
Period: Overall Study
Arm/Group | MORAb-009 Plus Gemcitabine ('MORAb-009') | Placebo Plus Gemcitabine ('Placebo')
Started | 78 | 77
Completed | 0 | 0
Not Completed | 78 | 77
Not completed — Adverse Event | 16 | 9
Not completed — Death | 7 | 7
Not completed — Lack of Efficacy | 40 | 49
Not completed — Physician Decision | 2 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Discontinuation of Study by the Sponsor | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MORAb-009 Plus Gemcitabine ('MORAb-009') | Placebo Plus Gemcitabine ('Placebo') | Total
Number analyzed (Participants) | 78 | 77 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 77 | 155
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (12.7) | 65.8 (10.3) | 65.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 77
  Male | 39 | 39 | 78
Race/Ethnicity, Customized [Number; unit: Participants]
  African American | 2 | 2 | 4
  Asian | 0 | 3 | 3
  Hispanic | 6 | 4 | 10
  White - White/Caucasian/European Heritage | 69 | 67 | 136
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  North America | 57 | 57 | 114
  Europe | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: This measure was defined as the time (in months) from the date of randomization to the date of death, whatever the cause. The primary endpoint was analyzed when 110 events (deaths) were observed. In the absence of death confirmation or for subjects alive at the time of analysis, the survival time will be censored at the date of the last study follow-up.
Time Frame: 1-21 Months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MORAb-009 Plus Gemcitabine ('MORAb-009') | Placebo Plus Gemcitabine ('Placebo')
Number analyzed (Participants) | 78 | 77
Months | 6.5 [4.5 to 8.10] | 6.9 [5.4 to 8.8]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free Survival (PFS) is defined as the time from the date of randomization to the date of the first observation of disease progression (clinical or radiological) or death due to any cause. Progression is defined, using RECIST, as a measurable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline. If progression or death is not observed, the PFS time will be censored at the date of the last tumor assessment without evidence of progression prior to the date of initiation of further anticancer treatment.
Time Frame: 1-21 Months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MORAb-009 Plus Gemcitabine ('MORAb-009') | Placebo Plus Gemcitabine ('Placebo')
Number analyzed (Participants) | 78 | 77
Months | 3.4 [1.9 to 4.7] | 3.5 [2.8 to 4.9]

3. Secondary Outcome: Best Overall Response Rate
Description: Best overall response is the number of participants with a Complete Response (CR) or Partial Response (PR), as classified by independent blinded review of the CT or MRI images, based on RECIST 1.0. A CR is the disappearance of all target lesions. PR is at least a 30% decrease in the sum of the longest diameters of target lesions, taking as a reference the baseline sum longest diameter. Progressive Disease (PD) is at least a 20% increase in the sum of the longest diameters of target lesions or the appearance of one or more new lesions. Stable disease (SD) is neither CR, PR or PD.
Time Frame: Baseline to response up to 21 months
Measure: Number; unit: percentage of participants
Arm/Group | MORAb-009 Plus Gemcitabine ('MORAb-009') | Placebo Plus Gemcitabine ('Placebo')
Number analyzed (Participants) | 78 | 77
percentage of participants
  Complete or Partial Response | 6.4 | 7.8
  Complete Response | 0 | 0
  Partial Response | 6.4 | 7.8
  Stable Disease | 47.4 | 55.8
  Progressive Disease | 19.2 | 23.4
  Not Evaluable | 26.9 | 13.0

ADVERSE EVENTS:
Time Frame: From Baseline up to 21 months.
Description: 73 participants received MORAB-009 plus gemcitabine and 75 participants received Placebo plus gemcitabine.
Arm/Group | MORAb-009 Plus Gemcitabine ('MORAb-009') | Placebo Plus Gemcitabine ('Placebo')
Serious Adverse Events (participants affected / at risk) | 49/73 | 54/75
Other Adverse Events (participants affected / at risk) | 73/73 | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-009 Plus Gemcitabine ('MORAb-009') (N=73) | Placebo Plus Gemcitabine ('Placebo') (N=75)
Vomiting (Gastrointestinal disorders) | 6 | 6
Nausea (Gastrointestinal disorders) | 4 | 3
Abdominal Pain (Gastrointestinal disorders) | 3 | 3
Obstruction gastric (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 11
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 3
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 4
Cellulitis (Infections and infestations) | 1 | 4
Bacteremia (Infections and infestations) | 0 | 4
Sepsis (Infections and infestations) | 2 | 1
Abdominal Abscess (Infections and infestations) | 0 | 1
Biliary Sepsis (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthenia (General disorders) | 4 | 1
General physical health deterioration (General disorders) | 1 | 4
Pyrexia (General disorders) | 2 | 3
Chest pain (General disorders) | 0 | 2
Generalized oedema (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 7
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Poor venous access (Vascular disorders) | 1 | 0
Thromboangiitis obliterans (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Nephritis (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
International normalized ratio increased (Investigations) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Parenteral nutrition (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-009 Plus Gemcitabine ('MORAb-009') (N=73) | Placebo Plus Gemcitabine ('Placebo') (N=75)
Nausea (Gastrointestinal disorders) | 35 | 38
Constipation (Gastrointestinal disorders) | 34 | 27
Abdominal pain (Gastrointestinal disorders) | 27 | 20
Vomiting (Gastrointestinal disorders) | 23 | 24
Diarrhoea (Gastrointestinal disorders) | 22 | 23
Abdominal distention (Gastrointestinal disorders) | 12 | 10
Abdominal pain upper (Gastrointestinal disorders) | 3 | 11
Ascites (Gastrointestinal disorders) | 8 | 5
Flatulence (Gastrointestinal disorders) | 9 | 4
Dyspepsia (Gastrointestinal disorders) | 7 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 5
Fatigue (General disorders) | 32 | 32
Oedema peripheral (General disorders) | 27 | 23
Pyrexia (General disorders) | 13 | 26
Asthenia (General disorders) | 15 | 18
Chills (General disorders) | 13 | 14
Oedema (General disorders) | 6 | 4
Pain (General disorders) | 2 | 7
Chest pain (General disorders) | 4 | 3
General physical health deterioration (General disorders) | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 26 | 25
Dehydration (Metabolism and nutrition disorders) | 13 | 15
Hypokalemia (Metabolism and nutrition disorders) | 12 | 13
Hyponatremia (Metabolism and nutrition disorders) | 7 | 6
Decreased appetite (Metabolism and nutrition disorders) | 3 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 2
Anaemia (Blood and lymphatic system disorders) | 32 | 36
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 25
Neutropenia (Blood and lymphatic system disorders) | 16 | 20
Leukopenia (Blood and lymphatic system disorders) | 11 | 16
Weight decreased (Investigations) | 10 | 9
Blood alkaline Phosphatase increased (Investigations) | 9 | 8
Alanine aminotransferase increased (Investigations) | 8 | 6
Aspartate aminotransferase increased (Investigations) | 8 | 5
Neutrophil count decreased (Investigations) | 5 | 6
Haemoglobin decreased (Investigations) | 7 | 3
Blood bilirubin increased (Investigations) | 4 | 5
Platelet count decreased (Investigations) | 3 | 6
International normalised ratio increased (Investigations) | 6 | 2
Urinary tract infection (Infections and infestations) | 12 | 10
Cellulitis (Infections and infestations) | 5 | 8
Pneumonia (Infections and infestations) | 4 | 5
Candidiasis (Infections and infestations) | 3 | 4
Rhinitis (Infections and infestations) | 2 | 4
Bacteraemia (Infections and infestations) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 11 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 6
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 11
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Dizziness (Nervous system disorders) | 12 | 12
Headache (Nervous system disorders) | 7 | 9
Dysgeusia (Nervous system disorders) | 6 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 5
Deep vein thrombosis (Vascular disorders) | 7 | 11
Hypertension (Vascular disorders) | 5 | 10
Hypotension (Vascular disorders) | 5 | 6
Pallor (Vascular disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 13 | 10
Anxiety (Psychiatric disorders) | 8 | 6
Depression (Psychiatric disorders) | 4 | 5
Sleep disorder (Psychiatric disorders) | 2 | 5
Confusional state (Psychiatric disorders) | 5 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 8
Cholangitis (Hepatobiliary disorders) | 2 | 4
Jaundice (Hepatobiliary disorders) | 2 | 4
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 11
Palpitations (Cardiac disorders) | 4 | 2
Tachycardia (Cardiac disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less